CLINICAL TRIAL: NCT06117345
Title: Enhancing Parent/Caregiver Engagement in the Pediatric Intensive Care Unit (PICU): A Pilot Study of a PICU Journal Intervention
Brief Title: Enhancing Parent/Caregiver Engagement in the Pediatric Intensive Care Unit (PICU): A PICU Journal
Acronym: PICUJournal
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Jessika Boles, Co-PI, Vanderbilt University Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 231386
Record Dates: First submitted 2023-10-23; First posted 2023-11-07 (Actual); Last update posted 2025-06-02 (Actual); Status verified 2025-05

CONDITIONS: Critical Illness
Keywords: Critical care; Intensive care; Pediatrics; Family-Centered Care; Family Engagement; PICU Liberation
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Parents/Caregivers (Experimental): Parents/caregivers of children hospitalized in the PICU at Monroe Carell Jr. Children's Hospital at Vanderbilt who will participate in the PICU journal intervention
  Interventions: Behavioral: PICU Journal
- Patients (No Intervention): Pediatric patients ages 8 to 18 years whose parents/caregivers participated in the PICU journal intervention
- PICU providers and staff (No Intervention): PICU providers and staff who observed or participated in the PICU journal intervention during its use with parents/caregivers

INTERVENTIONS:
Behavioral: PICU Journal — A hard-copy, customizable educational/therapeutic/expressive journal for parents/caregivers to seek information and document their child's PICU experiences and outcomes.
  Other Names: PICU diary
  Arms: Parents/Caregivers

SUMMARY:
Admission to the pediatric intensive care unit (PICU) is well-recognized to be extremely distressing and stressful for the patient and family. As medical research and technology have advanced more and more children in the PICU are surviving, however in turn incurring new and persistent impairments across physical, cognitive, emotional, and social domains of health. This phenomenon is often referred to as post-intensive care syndrome (PICS). These impairments not only impact the patient but parents have also been found to have poor emotional health outcomes following discharge from the PICU.

Consistently, parents/caregivers of children admitted to the PICU report their primary concerns to be 1) the overwhelming physical environment of the PICU, 2) uncertainty about the child's survivorship and outcomes, 3) relationships and communication with staff, and 4) feeling helpless. Additionally, research has shown that caregiver-perceived stress during the child's hospitalization positively predicts post-traumatic stress three months after discharge for parents/caregivers (Nelson et al., 2019), which may translate into higher risk and duration of post-traumatic stress in their children. Therefore, providing an in-hospital outlet such as a "PICU Journal" for patients and families to express their subjective experiences may help bridge the gap between perception and reality as a means of buffering against post-traumatic responses. Conceptually, a semi-structured journal intervention may integrate the therapeutic aspects of journaling while also providing pertinent information and serving as an advocacy and communication tool. Prior research has demonstrated the use of a "PICU Journal" is feasible for implementation and has been well-received by families of children in the PICU (Herrup et al., 2019).

Therefore, the aims of this mixed-method study are to 1) examine the relationship between this journaling intervention and the perceived stress, care engagement, symptoms of anxiety, and depression, and the development of PICS in parents of children hospitalized in the PICU, and 2) examine the relationship between parent participation in this intervention and the development of PICS-p in children, and 3) assess the feasibility of this intervention from key stakeholders.

DETAILED DESCRIPTION:
Eligible participants will be identified by their primary Certified Child Life Specialist (CCLS) using the daily PICU census and electronic medical record. All eligible participants will first be approached by the child life specialist on their care team to provide brief information about the study and refer to the key study personnel (KSP) if the parent/caregiver is interested in learning more. If they are potentially interested in participating, a member of the KSP (comprised of a doctoral level CCLS, psychology graduate students, PICU physician, and research nurses) will approach the parent/caregiver at bedside and give information and obtain consent. When approaching for consent, the KSP will first obtain approval to approach from the patient's bedside nurse to ensure it is a feasible and appropriate time to do so. All parents/caregivers who indicate interest will be approached to participate to ensure a diverse and broad sample, until a total of 75 parents/caregivers have completed participation in the study. No randomization will be used.

Once consent has been given by the parent/caregiver (using an electronic consent form housed in REDCap), they will complete a short demographic survey in REDCap. The family will then be given the PICU Journal along with supplies and instructions on how to access additional pages and the photo printer. The PICU Journal was developed by conducting extensive research on perceived stressors in the PICU, post-intensive care syndrome in pediatrics and their families, and the use of dairies in the intensive care unit setting, along with consultation from Certified Child Life Specialists, and with input from family advisors. Families will be able to take the original journal home with them.

Data will be collected at three-time points: time one (T1) between 24 and 72 hours of the child's admission, time two (T2), peri-discharge, and time three (T3) three months post-discharge.

Timepoint 1 (T1) Between 24 - 72 hours after admission:

Parent Participation Consent Form Illness Severity (Chart Review) Child Demographics (Chart Review) Parent Demographics Survey Abbreviated Parental Stressor Scale: Pediatric Intensive Care Unit (APSS: PICU) Caregiving Health Engagement Scale (CHE-s)

Timepoint 2 (T2) Peri-discharge Abbreviated Parental Stressor Scale: Pediatric Intensive Care Unit (A-PSS: PICU) Caregiving Health Engagement Scale (CHE-s) Hospital Anxiety and Depression Scale (HADS) Journal Use & Satisfaction Survey

Timepoint 3 (T3) 3 months post-discharge:

Hospital Anxiety and Depression Scale (HADS) Impact of Events Scale-Revised (IES-R) At Home Journal Use & Satisfaction Survey Child Participation Assent Form (Child Report) Child Revised Impact of Events Scale (CRIES-8) (Child Report)

*Semi-Structured Interview (Parents)

At the conclusion of the study :

Provider Satisfaction Survey

ELIGIBILITY:
Parent/Caregiver Inclusion Criteria:

* The participant is a primary caregiver of a pediatric patient (ages 1 month to 21 years) admitted to the pediatric intensive care unit (PICU) at Monroe Carell Jr. Children's Hospital at Vanderbilt (MCJCHV)
* The participant's child meets the criteria for Levels 1 or 2 of the Early Mobility Protocol at MCJCHV
* The participant's child has been hospitalized in the PICU for between 24 and 72 hours at the time of informed consent.
* The participant has not had prior experience with their child(ren) being admitted to the PICU.
* The participant is proficient in reading and writing the English language.

Parent/Caregiver Exclusion Criteria:

* The participant is unwilling to provide consent.
* The participant is unable to read and write in the English language.

Child Inclusion Criteria:

* The child participant is between the ages of 8 to 17 years.
* The participant is proficient in reading and writing the English language.

Child Exclusion Criteria:

* The participant is unwilling to provide assent.
* The participant is unable to read and write in the English language.

Staff Inclusion Criteria:

* The participant(s) interact with patients in the PICU at Monroe Carell Jr. Children's Hospital at Vanderbilt.
* The participant is proficient in reading and writing the English language.

Staff Exclusion Criteria

- The participant is unable to read and write in the English language.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2026-07-15 (Estimated); Study Completion 2026-11-15 (Estimated)

PRIMARY OUTCOMES:
Parent/Caregiver reported stress level | At study enrollment (T1), within 48 hours of child's discharge from hospital (T2)
  Score on the Abbreviated Parental Stressor Scale: Pediatric Intensive Care Unit; 7 Likert type items scored from 1 to 5, with 1 being "not stressful" and 5 being "extremely stressful." Composite scores can range from 0 (not experienced) to 35 (extremely stressful).
Parent/Caregiver care engagement level | At study enrollment (T1), within 48 hours of child's discharge from hospital (T2)
  Score on the Caregiving Health Engagement Scale; 7 items with four answer choices scored from 1 to 4. Composite scores can range from 7 (minimal engagement) to 28 (high engagement).
Parent/Caregiver reported depression and anxiety symptoms | within 48 hours of child's discharge from hospital (T2), at 3 months post-discharge (T3)
  Score on the Hospital Anxiety and Depression Scale; two subscales (anxiety and depression) with 7 items each. Items have 4 answer choices scored from 1 to 4, with higher numbers indicating higher alignment with anxiety or depression. Cut scores are used to determine clinical significance; a total score of less than 7 on a subscale indicates a non-case, 8-10 on a subscale indicates mild, 11-14 indicates moderate, and 15 to 21 is considered severe.
Parent/caregiver reported impact of events | at 3 months post-discharge (T3)
  Score on Impact of Events Scale-Revised; 20 Likert-type items scored from 0 (not experienced) to 4 (extremely distressed). Total composite scores can range from 0 (not experienced) to 80 (extremely distressed).
Parent/Caregiver use of and satisfaction with PICU journal | within 48 hours of child's discharge from hospital (T2), at 3 months post-discharge (T3)
  Responses to a descriptive survey created by research team to assess frequency/type of PICU journal use and completion, as well as parent/caregiver perceptions of feasibility and utility
Child reported impact of events | at 3 months post-discharge (T3)
  Score on the Child Revised Impact of Events Scale; 8 items with four answer choices scored from 0 (not at all) to 3 (often). Total composite scores can range from 0 (not at all distressed) t to 24 (extremely distressed).
Parent/caregiver Experiences Interview | at 3 months post-discharge (T3)
  Responses to semi-structured interview about PICU journal perceptions and experiences (in-person, by phone, or by teleconference)
PICU Staff perceptions of PICU journal intervention | Through study completion, an expected average of 2 years
  Responses to a descriptive survey created by research team to collect perceptions about and level of engagement with PICU journal intervention

CONTACTS AND LOCATIONS:
Overall Officials: Kristina Betters, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Monroe Carell Jr. Children's Hospital at Vanderbilt, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No